CLINICAL TRIAL: NCT04590651
Title: Cataract Surgery in Patients With Pseudoexfoliation and Pseudoexfoliation Glaucoma
Acronym: PHACOPXG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peeter Kuddu (Other)
Responsible Party: Sponsor-Investigator, Peeter Kuddu, Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHACOPXG
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Pseudoexfoliation; Pseudoexfoliation Syndrome; Pseudoexfoliation Glaucoma; Cataract
MeSH Terms: conditions — Exfoliation Syndrome; Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient will not know which group he or she has been randomised to during the duration of the study. The care provider and investigator will not know the randomisation before the patient is enrolled in the study. The care provider and investigator will know the randomisation group at the time of randomisation, which will take place after the preoperative data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PHACO cataract surgery (Experimental): In this group normal phacoemulsification cataract surgery will be preformed.
  Interventions: Procedure: Cataract surgery
- PHACO + extra aspiration (Experimental): In this group an extra one minute anterior chamber angle aspiration will be preformed at the end of a standard cataract operation.
  Interventions: Procedure: Cataract surgery with extra anterior chamber angle aspiration

INTERVENTIONS:
Procedure: Cataract surgery — Routine phacoemulsification cataract surgery using the Alcon Centurion® device.
  Other Names: Phacoemulsification
  Arms: Standard PHACO cataract surgery
Procedure: Cataract surgery with extra anterior chamber angle aspiration — Routine phacoemulsification cataract surgery using the Alcon Centurion® device. At the end of the case a one minute extra anterior chamber angle aspiration will be preformed after the removal of the viscoelastic agent.
  Other Names: Phacoemulsification with extra anterior chamber angle aspiration
  Arms: PHACO + extra aspiration

SUMMARY:
The study aims to document the effect cataract surgery has on the pseudoexfoliation and pseudoexfoliation glaucoma eye. Details such has patient history, history of possible glaucoma, intraocular pressure, status of the eye, operation parameters and postoperative effect will be documented. The study is prospective and randomised . Patients will be divided in to two groups: in one standard phacoemulsification cataract surgery will be preformed. In the second group the anterior chamber angel will be aspirated an extra minute at the end of the case with the IA probe. The aim is to determine weather this extra aspiration will have an effect on postoperative intraocular pressure and other parameters.

DETAILED DESCRIPTION:
This randomized clinical trial will be performed at the Helsinki University Central Hospital. Patients that are eligible for cataract surgery will be recruited. A history of pseudoexfoliation or pseudoexfoliation glaucoma is required.

Preoperative data such as age, sex, ethnicity, history of diabetes and history of high blood are recorded. If the participant has pseudoexfoliation glaucoma the following data will be recorded: number of years elapsed since the diagnosis; number of glaucoma medications; number of active agents; possible bilateral disease.

Visual acuity is attained during every visit (preoperatively and 1 day, 1 week, 1 month, 6 months, 1 year, 2 years and 3 years postoperatively) using the Snellen chart. Both uncorrected and best corrected visual acuity are attained.

Intraocular pressure (IOP) is also attained during every visit using the Goldmann applanation tonometer (measured twice during each visit). The measurements will be taken between 8 a.m and 12 p.m to minimize the effect of diurnal fluctuations.

Biomicroscopy will be done preoperatively to assess the following: conjunctival hyperemia; possible pseudoxfoliation material on the endothelium, iris border and lens capsule; anterior chamber angle opening (grade 0-4 using the Shaffer system); existence of the Sampaolesi line; iris dilatation in millimeters (20 minutes after instilling 1 drop of tropicamid 5mg/ml and 1 drop of 2,5% phenylephrine; nuclear sclerosis (grades 0-4); presence of phacodonesis.

Postoperatively the anterior chamber is assessed for inflammation using the SUN nomenclature at 1 day, 1 week, 1 months and 6 months.

Preoperatively axial length (AL), anterior chamber depth (ACD) and lens thickness (LT) are obtained using the Haag-Streit LensStar optical biometer. Lens calculations are done using the SRK/T, Hoffer Q, Holladay II and Barrett formulas and the best suited IOL determined.

Anterior chamber OCT (Tomey Casia 2) is attained preoperatively and at at 1 months, 6 months and 1 year postoperatively. The following parameters are recorded: angle opening distance (AOD) and trabecular iris surface area (TISA). Both at 500 and 750 micrometers. Nasal and temporal (0 and 180 degrees) sites will be analyzed.

Specular microscopy will be performed preoperatively and 1 year postoperatively using the Konan CellChek device. Cell density (cells per mm2) will be evaluated.

Macular OCT using the Heidelber Spectralis device is attained preoperatively and one month postoperatively. The central retinal thickness (CRT) will be documented. The vitreoretinal surface and Bruch's membrane are used as measuring points.

The ocular nerve head OCT obtained using the Heidelberg Spectralis OCT. The global nerve fiber layer thickness is documented preoperatively, and possible progression is assessed by a glaucoma specialist (NL) at 1 month, 1 year, 2 years and 3 years postoperatively.

The Kona FM-600 cell flare meter is also used to assess inflammation preoperatively and at 1 day, 1 week, 1 month, 6 months and 1 year postoperatively.

The visual field will be analyzed using the Haag-Streit Octopus static perimeter with the G program. Perimetry is performed at 1 month ,1 year, 2 years and 3 years postoperatively. Mean defect (MD), square root of loss variance (sLV) and reliability factor will be documented.

Randomisation is done before the cataract surgery after the preoperative evaluation. Stratified block randomization is used to ensure that intraocular pressure and participant age do not vary too much between the groups. The participants are randomized into two groups: in the first group standard phacoemulsification is performed and an intraocular lens (IOL) is implanted. In the second group an extra one-minute anterior chamber angle aspiration is preformed using the IA tip after all the viscoelastic is aspirated from the anterior chamber. The aim is not to touch the chamber angle with the IA tip but rather make continuous sweeping motions under visual control during that minute.

Three surgeons (KK; ML; PK) from the Department of Corneal and Anterior Segment Surgery are designated to perform the surgeries. Preoperative drops include one drop of tropicamide 5 mg/ml, 2,5% phenylephrine and apraclonidine 10 gm/ml. The eye is disinfected with either iodine or chlorhexidine drops, and the lids swiped with alcohol swabs. XylocainⓇ 2% gel is used for anesthetic after rinsing the surface of the globe. The main incision is 2,4 mm and the side port 1 mm wide. Intracameral lidocaine and phenylephrine are used after making the side port incision. DiscoViscⓇ and ViscoatⓇ can be used as viscoelastic agents during surgery. The use of a Malyugin ring Ⓡ , iris hooks, capsular support hooks and a capsular tension ring is permitted. The need for these instruments will be determined by the surgeon during the procedure. Phacoemulsification is performed using the stop & chop or direct chop technique. The Alcon CenturionⓇ device is used in all surgeries with the same predetermined settings. Johnson & Johnson TecnisⓇ monofocal 1-piece IOL (ZCB00) is used in all cases. The following data is recorded during surgery: surgeons initials; surgery time in minutes (form the time the first incision is made to the time the wounds are sealed); surgery technique; the use of a Malyugin Ⓡ ring or capsular tension ring; the use of iris hooks or capsular support hooks; cumulative dissipated energy (CDE); ultrasound total time; total aspiration time; estimated fluid aspirated; fluid used ( calculated by subtracting the amount of fluid left at the end of the case form the amount left after priming the phaco device); possible extra anterior chamber angle aspiration.

Postoperatively a drop of apraclonidine 10 mg/ml is instilled after a 30 to 60-minute period of monitoring the patient in the recovery room. If the intraocular pressure pressure is under 5 or over 25 (measured with the iCareⓇ rebound tonometer by a nurse) the surgeon is asked to assess the situation.

Complications such as posterior capsule rupture and suprachoroidal hemorrhage are grounds for discontinuation of participation in the study.

The postoperative visits take place at 1 day, 1 week, 1 month, 6 months, 1 year, 2 years and 3 years. The types of examinations preformed are described in detail above.

The primary aim of this study is to determine the change in intraocular pressure postoperatively. The study also aims to determine the factors effecting the change in IOP. For this reason, patient history, glaucoma history, the status of the eye and data form the surgery are recorded and numerous tests will be performed. These are described in detail above. This study is aimed to aid clinicians in everyday work, for that and safety reasons a wash-out period will not be included. Adding additional glaucoma medication is permitted during the course of the study and the number of medications and active agents is documented during the postoperative exams. The need for additional glaucoma medication will be assessed during follow-up examinations with the aid of IOP measurement, ONH-OCT and perimetry.

The study also aims to determine the rate of macular edema at 1 month postoperatively, for that reason the central retinal thickness is recorded preoperatively and at 1 month postoperatively using the Heidelberg Spectralis OCT device.

The study will also determine the rate of endothelial cell loss at 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The patient has to meet the criteria set by the Helsinki Central University hospital for cataract surgery: best corrected visual acuity of 0,5 (Snellen) or below in the better eye or 0,3 (Snellen) or below in the worse eye; glare or other debilitating symptoms determined to be caused by cataract; cataract interfering with the diagnosis or follow up of glaucoma
* Pseudoexfoliation or pseudoexfoliation glaucoma

Exclusion Criteria:

* Previous intraocular surgery of any kind
* Previous glaucoma surgery or cyclophotocoagulation
* Previous selective laser trabeculoplasty (SLT) or argon laser trabeculoplasty (ALT)
* Any other ocular pathology likely to demand surgery during the course of the study
* Wet age related macular degeneration (wetAMD)
* Need for glaucoma surgery determined by a glaucoma specialist in cases where the intraocular pressure is deemed to high compared to the ocular nerve head condition and/or visual field defect.
* History of uveitis.
* History of herpetic keratitis.
* History of ocular trauma.
* Dementia or other conditions preventing the patient from adhering to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-06-11 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
IOP Change | IOP will be measured preoperatively and at 1 day, 1 week, 1 month, 6 months, 1 year, 2 years and 3 years postoperatively.
  Intraocular pressure (IOP) measured twice during every visit with a Goldmann applanation. tonometer. Measurements will be taken before 12 p.m local time. Change from baseline is being measured at these specified times.

SECONDARY OUTCOMES:
Visual acuity change | Preoperative and at 1 day, 1 week, 1 month, 6 months, 1 year, 2 years and 3 years postoperatively.
  Uncorrected and best corrected visual acuity will be documented during every visit using the Snellen visual acuity chart. Change from baseline is being measured at these specified times.

OTHER OUTCOMES:
Inflammation change | Measured preoperatively and at 1 day, 1 week, 1 month, 6 months and 1 year postoperatively.
  Measured with the the Kona FM-600 flare meter. Photon count per millisecond. Change from baseline is being measured at these specified times.
Cell density change | Measured preoperatively and 1 year after surgery
  Endothelial cell density measured with the Konan CellChek specular microscope. Cell count per mm2. Change from baseline is being measured at these specified times.
Central retinal thickness change | Preoperatively and at 1 month postoperatively.
  Central retinal thickness is measured by the Hidelberg Spectralis OCT. Measured in micrometers. The distance between the pigment epithelium and internal limiting membrane. Change from baseline is being measured at these specified times.
ONH-OCT change | Measured preoperatively and at 1 month, 6 months, 1 year, 2 years and 3 years postoperatively.
  Ocular nerve head OCT. Measured with the Heidelberg Spectralis OCT. Possible thinning of the nerve fiber layer determined by a glaucoma specialist (NL). Change from baseline is being measured at these specified times.
Visual Field change | Measured 1 month, 1 year, 2 years and 3 years postoperatively.
  Visual Field measured with Haag-Streit Octopus static perimeter. The G program is used. Change from baseline is being measured at these specified times.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Krootila, AP, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After the conclusion of the study for 2 years
Access Criteria: Access granted for healthcare professionals, investigators and the peer-review process.